CLINICAL TRIAL: NCT01626560
Title: Effects of Daptomycin in the Levels of IL-1, IL-6 and TNF in Patients With Complicated Cellulitis/Erisipela in Comparison With Vancomycin or Oxacillin
Brief Title: The Effects of Daptomycin and Cytokines Production in Comparison With Vancomycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Evangelico de Curitiba (Other)
Responsible Party: Principal Investigator, Felipe Francisco Bondan Tuon, PhD, Hospital Universitario Evangelico de Curitiba
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: daptocina
Record Dates: First submitted 2012-03-23; First posted 2012-06-22 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomicina (Other)
  Interventions: Drug: Daptomycin
- Vancomycin (Other)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Daptomycin — daptomycin 4-6mg/kg qd 10 - 14 days
  Arms: Daptomicina
Drug: Vancomycin — Vancomycin 1g q12h 10 - 14 days
  Arms: Vancomycin

SUMMARY:
Primary: To determine the influence of daptomycin on inflammatory cytokine (IL-1, TNF and IL-6) for the treatment of complicated cellulitis/erysipela compared with alternative treatment (vancomycin or oxacillin). Secondary: To evaluate the clinical outcome of both groups according to levels of the cytokines evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients will be age between 18 and 65 who required hospitalization and parenteral antimicrobial therapy
2. Clinical documentation of cellulitis / erysipela
3. Documentation of a minimal surface area 75 cm2 based on the length and / or width of the redness, swelling and / or induration
4. Documented fever, defined as oral or tympanic temperature greater than or equal to 38 ° C

Exclusion Criteria:

1. Infections and other minor addition of erysipelas / cellulitis
2. Any recent use of antibacterial drug therapy (systemic or topical antibacterial drugs within 14 days of enrollment)
3. Patients with clinical conditions that alter the interpretation of the primary outcome as patients with neutropenia or compromised immune function, as HIV infection, autoimmune disorders, use of corticosteroids.
4. Patients with known or suspected osteomyelitis.
5. Patients with suspected or confirmed septic arthritis.
6. Patients with complicated skin infections, such as diabetic foot infections. 7. Chronic use of antipyretic drugs (eg, daily use of naproxen).

8. Less than 18 years of age. 9. pregnancy 10. Patients with mixed infections of Gram-negative or be deleted since the therapy of gram-negative can influence the levels of cytokines.

11. Patients with renal clearance <30 mL / min. 12. Patients who are not susceptible to daptomycin or vancomycin. 13. Allergy to study medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cytokine levels | AUC will be calculated with multiple time points over a period of 14 days (0, 4, 8, 12 , 16, 24, 48, 72, 96, 120 and 168 hours post-dose)
  The results of cytokine levels will be evaluated after completion of antibiotic therapy, when testing will take place in the laboratory. Thus the measurement of cytokines will not be used to evaluate the clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Evangelico de Curitiba, Curitiba, Paraná, Brazil